CLINICAL TRIAL: NCT06568276
Title: The Benefit of Repairing the Deltoid Ligament in Unstable Ankle Fractures: Patient-reported Functional Outcome and Radiological Stability Measurements
Brief Title: The Benefit of Repairing the Deltoid Ligament in Unstable Ankle Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Sykehuset Innlandet HF (Other); Helse Nord-Trøndelag HF (Other); Helse-Bergen HF (Other); Norwegian Institute of Public Health (Other Government); Helse Stavanger HF (Other Government); Trondheim University Hospital (Other); Norwegian University of Science and Technology (Other); Alesund Hospital (Other); Nordlandssykehuset HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024104
Record Dates: First submitted 2024-05-22; First posted 2024-08-23 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Ankle Fractures; Deltoid Ligament; Sprain (Strain) (Ankle)
MeSH Terms: conditions — Ankle Fractures; Sprains and Strains

STUDY DESIGN:
Intervention Model Description: Multicentre Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (No Intervention): Unstable Weber B fractures receiving standard treatment, plate and screw fixation of the lateral malleolus only
- Additional deltoid ligament suture (Experimental): Unstable Weber B fractures receiving standard treatment, plate and screw fixation of the lateral malleolus and additional deep deltoid ligament suture
  Interventions: Procedure: Additional deep deltoid ligament suture

INTERVENTIONS:
Procedure: Additional deep deltoid ligament suture — The deep deltoid ligament will be sutured through a curved incision lifting the tibialis posterior tendon out to be sutured back after tying the ligament to an anchor in the talus.
  Arms: Additional deltoid ligament suture

SUMMARY:
Ankle fractures occur in 1 out of 800 persons a year and is a common injury. The deltoid ligament is necessary for the stability of the joint and guides choice of treatment. Cadaveric studies have shown that deltoid ligament repair gives more stability than the osteosynthesis of the lateral malleolus itself. The investigators want to show if suture of the deltoid ligament in unstable ankle fractures contribute to a better functional result and/or prevent long term osteoarthritis for our participants. Patients sustaining severe ankle fractures have shown a considerable loss of function that might affect their long term activities of daily living (ADL) function. Improving outcome for this group may preserve some patients' ability to work and reduce community expenses.

DETAILED DESCRIPTION:
During the last two decades less severe ankle fractures have been shown not to need operative treatment in general. The total number of ankle fracture surgeries has gone down. Therefore, surgically treated ankle fractures nowadays are on average more complex. The understanding of these injuries implies a recognition of the role of the deep deltoid ligament as a main stabilizer of the ankle joint. Deltoid ligament repair is documented to be a good option to regain ankle joint anatomy from smaller studies. This repair also compensates for syndesmotic injury to some extent. The effect of deep deltoid ligament repair in Weber B ankle fractures and its effect on long term function and arthritis is not yet known from clinical studies.

The investigators aim to show whether deltoid ligament suture gives a clinically significant superior result than solely osteosynthesis of the lateral malleolus in unstable ankle fractures. This will be performed as a multicentre randomized controlled study.

ELIGIBILITY:
Inclusion criteria; fluent in oral and written Norwegian language

* isolated Weber type B fractures and Weber B+ posterior malleolar Mason Molloy class I.
* Initial medial clear space (MCS)>=7mm or weightbearing x-ray evaluated as unstable or primary reposition after fracture dislocation.
* Pre-injury walking ability without aids.

Exclusion criteria

* assumed not compliant (drug use, cognitive- and/or psychiatric disorders).
* previous history of ipsilateral ankle fracture or ipsilateral major ankle-/foot surgery.
* open fx Gustilo Anderson II or more, multi-trauma and pathologic fracture.
* neuropathies and generalized joint disease such as Rheumatoid Arthritis or other more severe condition in same extremity
* fixation of tibial fragment or syndesmotic screw or suture button planned prior to surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2032-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient-reported functional outcome 1 year after injury | 1 and 2 years after injury, function 5 years after injury will also be collected
  Function will be measured in Olerud-Molander Ankle Score (OMAS) (ankle specific) (0 (worst)-100 (best))
Differences in radiological stability parameters with or without ligament suture at group level | 1 and 2 years after injury, function 5 years after injury will also be collected
  Differences in medial clear space (mm) on weightbearing x-rays or Gravity test at group level

SECONDARY OUTCOMES:
General health state reported through a general (generic) Patient-reported outcome measure (PROM) | up to 5 years
  The generic Euroquol EQ-5D (EQ 5D-5L) reports general health based on 5 items where Index scores range from -0.59 to 1; 1 is the best possible health state. Negative values represent health states perceived as worse than dead, which is equal to 0.
Posttraumatic ankle arthritis | 1,2 and 5 years
  Arthritis seen on weightbearing x-rays will be reported according to Kellgren Lawrence Scale (KGLS) (0 no arthritis to 4 severe/end stage arthritis with bone to bone contact and bone wear and osteophytes)
VAS Pain | 6 weeks, 3 months, 1, 2 and 5 years
  scale limited by intervals of no pain (0) and worst imaginable pain (100)
Patient-Reported Outcomes Measurement Information System (PROMIS) | 1, 2 and 5 years
  We will use a version of the Mobility bank 2.1. The setup and calculation method is still not clear. We await further progress from the organization developing this PROM. We hope to get a computer adapted testing (CAT) version of this survey ready in a Norwegian version within the start of 1 year follow up in September 2025
Self-reported Foot and Ankle Score (SEFAS) | 3 months, 1, 2 and 5 years
  Ankle specific PROM based on 12 items, scale 0(worst) - 48 (best possible)
Ankle Fracture Outcome of Rehabilitation Measure | 3 months, 1, 2 and 5 years
  Ankle Specific PROM based on 15 main items where 0 is the worst index score and 100 the best

OTHER OUTCOMES:
Complications | especially on first visits after surgery ie 6 and 12 weeks, and later visits up to 5 years after surgery.
  Infection, suture anchor malplacement, delayed/non-union and reoperation rate will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Frede Jon Frihagen, MD, PhD, Study Director — Oestfold Hospital Trust
Locations (9):
- Norway (9):
  - Oestfold Hospital Trust, Grålum, Postbox 300
  - Ålesund Sjukhehus, Ålesund
  - Haukeland University Hospital, Bergen
  - Nordlandssykehuset Bodø, Bodø
  - Sykehuset Innlandet Elverum, Elverum
  - Sykehuset Innlandet Gjøvik, Gjøvik
  - Sykehuset Levanger, Levanger
  - Oslo University Hospital Ullevål/Aker, Oslo
  - Stavanger University Hospital, Stavanger

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study protocol general august 2024 (2024-08-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT06568276/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: Study protocol update january 2025 (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT06568276/Prot_SAP_002.pdf